CLINICAL TRIAL: NCT06162429
Title: Comparison of Diagnostic Yield and Complication of Medical Thoracoscopy Using Flexible Bronchoscope Versus Semi-Rigid Pleuroscope Among Hospitalized Patients With Pleural Effusion
Brief Title: Medical Thoracoscopy With Flexible Bronchoscopy Versus Semi-Rigid Pleuroscope in Pleural Effusion (FLEXPLEUR)
Acronym: FLEXPLEUR
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Other Study IDs: FF-2023-128
Record Dates: First submitted 2023-11-19; First posted 2023-12-08 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flexible Thoracoscopy: Subjects with pleural effusion who underwent medical thoracoscopy using flexible bronchoscopy in the Respiratory Unit, Department of Internal Medicine, Faculty of Medicine UKM
  Interventions: Procedure: Flexible Bronchoscopy
- Semi-Rigid Pleuroscopy: Subjects with pleural effusion who underwent semi-rigid pleuroscopy using flexible bronchoscopy in the Respiratory Unit, Department of Internal Medicine, Faculty of Medicine UKM
  Interventions: Procedure: Semi-Rigid Pleuroscopy

INTERVENTIONS:
Procedure: Flexible Bronchoscopy — Subjects with pleural effusion who underwent medical thoracoscopy using flexible bronchoscopy
  Groups: Flexible Thoracoscopy
Procedure: Semi-Rigid Pleuroscopy — Subjects with pleural effusion who underwent medical thorascopy using semi-rigid pleuroscopy
  Groups: Semi-Rigid Pleuroscopy

SUMMARY:
Pleural effusion is a common problem in hospital patients. It may arise from a wide range of diseases. There is a multitude of recognised causes of pleural effusion, and in addition, other pleural conditions such as pleural thickening and pneumothorax represent a significant burden to the healthcare system and to patients. However, the diagnosis of this condition may sometimes be difficult. In pleural effusions undiagnosed by thoracocentesis, closed pleural biopsy increases the yield by ∼10% and 40%, respectively, in malignant and tuberculous pleural effusions, whereas the diagnostic yield of thoracoscopy is ∼93% in both malignant and tuberculous pleural effusions. Hence, medical thoracoscopy (MT) (pleuroscopy) is the gold standard in the diagnosis of pleural effusion and it is indicated when less invasive tests have failed. MT is a procedure in which the pleura is directly and visually examined. An endoscope is inserted into the intercostal space by creating a pneumothorax with an incision through the chest wall. The pleural space and its lining can be inspected and therapeutic interventions performed.

There are two different techniques that can be performed for diagnostic and therapeutic thoracoscopy. One method recommends a single-entry site, the use of a usually 9-mm rigid thoracoscope (or of a semi-rigid/semi-flexible 7-mm pleuroscope) with a working channel for accessory instruments and an optical biopsy forceps, both performed under local anaesthesia. The other method requires two entry sites: one for a 7-mm trocar for the examination telescope, and the other for a 5-mm trocar for accessory instruments including the biopsy forceps, and is usually performed with conscious sedation or general anaesthesia.

In the trained hands of a pulmonologist, MT is a safe and effective procedure for diagnosing and treating multiple pleural diseases. Valsecchi et al reported a pathological diagnostic yield of 71% over a span of 30 years in around 2000 patients. The unfamiliarity of the pulmonary physician with the rigid instrument and familiarity with the flexible bronchoscope has led various investigators to attempt thoracoscopy even with a fibreoptic bronchoscope.

The use of a flexible fibreoptic instrument to examine the pleural space was reported by Senno et al in the 1970s in the United States. Studies showed that flexible bronchoscope, when used as a thoracoscope, maintains a clear optical field by allowing concurrent suctioning, which is analogous to the suction techniques used during flexible bronchoscopy and better views at the apex and paravertebral gutters.This method is, therefore, considered to be useful for surgeons or physicians with experience in chest drainage and flexible bronchoscopy as well as safe and well tolerated with a minimal degree of discomfort and expense.

DETAILED DESCRIPTION:
RESEARCH QUESTION Can Medical thorascopy using a flexible bronchoscope be used as an alternative method to a semi-rigid pleuroscopy for diagnosis of pleural effusion with a comparable outcome?

RESEARCH HYPOTHESES

1. No difference in the diagnostic yield between flexible bronchoscopy and semi-rigid pleuroscopy
2. No difference in the complication rate between flexible bronchoscopy and semi-rigid pleuroscopy
3. Duration of procedure in flexible bronchoscopy is longer compared to semi-rigid pleuroscopy.
4. The predictors of diagnostic yield in flexible bronchoscopy are similar to semi-rigid pleroscopy.
5. No difeference in the specimen size taken from flexible bronchoscopy versus semi-rigid pleuroscopy

NOVELTY This is first study in Malaysia that we know of that has attempted to evaluate the diagnostic yield of medical thoracosopy using flexible bronchoscope and its complications. This study may be used to see whether there is a suitable alternative for respiratory physician to safely diagnosed pleural disease after a failed non-invasive procedure. While conventional medical thoracoscopy is the more expensive procedure, the true difference in procedure-related costs associated with flexible bronchoscope compared to semi-rigid pleuroscope is unknown due to the lack of cost-analysis study. Perhaps this study can provide the basis for future study to analyse the true cost-benefit of using flexible bronchoscope in medical thoracoscopy.

RESEARCH OBJECTIVES

GENERAL OBJECTIVE To compare the diagnostic yield, complication and duration of MT using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.

SPECIFIC OBJECTIVES

1. To compare the type of complication using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.
2. To compare the rate of complication using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.
3. To compare the duration of procedure using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.
4. To determine the predictors of diagnostic yield of flexible bronchoscope in hospital patients with pleural effusion.
5. To compare the size of biopsy samples from flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.

SIGNIFICANCE OF RESEARCH This research proposal is important to improve the diagnosis of hospital patients presenting with pleural effusion in Malaysia. Semi-rigid pleuroscope is expensive and not widely available, whereas flexible bronchoscope is more readily available and can be used as an alternative for medical thoracoscopic pleural biopsy. There is no previous study looking at diagnostic yield comparison between flexible bronchoscope and semi-rigid pleuroscope. This study could potentially serve as a feasibility study that can help future investigators prepare for full-scale research leading to intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Subjects admitted to Faculty of Medicine UKM during the study period and underwent a single MT with flexible bronchoscopy or semi-rigid pleuroscopy.

Exclusion Criteria:

1. Age < 18 years.
2. Patients with incomplete data
3. Patients' medical record that cannot be retrieved.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects admitted for pleural effusion who underwent a single MT with flexible bronchoscopy or semi-rigid pleuroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
To compare the diagnostic yield (in percentage) using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion. | between October 2017 to October 2022
  Subjects underwent medical thoracoscopy and the purpose is to compare the diagnostic yield, complication and duration of MT using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.

SECONDARY OUTCOMES:
To compare the rate of complication (in percentage) using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion. | between October 2017 to October 2022
  Subjects underwent medical thoracoscopy and the purpose is to compare the rate of complication using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.
To compare the duration of procedure (in minutes) using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion. | between October 2017 to October 2022
  Subjects underwent medical thoracoscopy and the purpose is to compare the duration of procedure using flexible bronchoscopy versus semi-rigid pleuroscopy in hospital patients with pleural effusion.
To determine the predictors of diagnostic yield of flexible bronchoscope in hospital patients with pleural effusion | between October 2017 to October 2022
  Subjects underwent medical thoracoscopy and the purpose is to determine the predictors of diagnostic yield of flexible bronchoscope in hospital patients with pleural effusion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, MBBS (IIUM), Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No